CLINICAL TRIAL: NCT04941807
Title: Use of Platelet-rich Plasma (PRP) Therapy in Patients With Brittle Nail Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Eclipse Aesthetics, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-07022437
Record Dates: First submitted 2021-06-21; First posted 2021-06-28 (Actual); Results first posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-03

CONDITIONS: Nail Diseases
Keywords: Nails; brittle nail syndrome; platelet-rich plasma
MeSH Terms: conditions — Nail Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Treatment is open-label with respect to patient and investigators but is blinded to an endpoint committee.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Platelet-rich plasma (Experimental): The proximal nail fold is cleansed with alcohol and platelet-rich plasma obtained from the patient is injected using a 1ml syringe and 30g needle, 0.1-0.2 ml of platelet-rich plasma is injected into 8 proximal nail folds.
  Interventions: Device: Platelet-rich plasma
- Platelet-poor plasma (Placebo Comparator): The proximal nail fold is cleansed with alcohol and platelet-poor plasma obtained from the patient is injected using a 1ml syringe and 30g needle, 0.1-0.2 ml of platelet-poor plasma is injected into 2 proximal nail folds.
  Interventions: Device: Platelet-poor plasma

INTERVENTIONS:
Device: Platelet-rich plasma — Blood will be drawn from a vein in the patient's arm into an 11 ml Eclipse platelet-rich plasma Tube. The blood is processed using a centrifuge machine from eclipse medical. After centrifugation, the platelet poor portion will be separated from the platelet-rich portion. The proximal nail folds are cleansed with alcohol. Using a 1ml syringe and 30g needle, 0.1-0.2 ml of platelet-rich plasma is injected into 8 proximal nail folds.
  Arms: Platelet-rich plasma
Device: Platelet-poor plasma — Blood will be drawn from a vein in the patient's arm into an 11 ml Eclipse platelet-rich plasma Tube. The blood is processed using a centrifuge machine from eclipse medical. After centrifugation, the platelet poor portion will be separated from the platelet-rich portion. The proximal nail folds are cleansed with alcohol. Using a 1ml syringe and 30g needle, 0.1-0.2 ml of platelet-poor plasma is injected into 2 proximal nail folds.
  Arms: Platelet-poor plasma

SUMMARY:
The purpose of this study is to assess the efficacy and safety of platelet-rich plasma therapy for brittle nail syndrome

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been diagnosed with brittle nails
* Must understand and voluntarily sign an informed consent form
* Must be male or female and aged 18-95 years at time of consent
* Must be able to adhere to the study visit schedule and other protocol requirements
* A nail clipping with histopathology that is negative for the presence of dermatophyte infection
* Patient must present with at least a score of 2 on the PGA scale.

Exclusion Criteria:

* Inability of the patient to provide written informed consent for any reason.

  * Subject has psoriasis, lichen planus, dermatophyte infection or other confounding abnormalities that are severe enough to result in a clinically abnormal fingernail
  * Use of any medication within 90 days prior to start of study
  * Inability to abstain for nail polishes, nail gels during the study period
  * Subject is pregnant or planning pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shari R Lipner, MD, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification.
Supporting Information: Study Protocol
Time Frame: Immediately following publication.
Access Criteria: Anyone who wishes to access the data.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from one location in the United States
Pre-assignment Details: A total of 11 participants passed screening and were randomized.
Units Other Than Participants: Fingernails
Period: Overall Study
Arm/Group | Platelet-rich Plasma | Platelet-poor Plasma
Started | 11; 80 Fingernails | 11; 22 Fingernails
Completed | 10; 73 Fingernails | 10; 20 Fingernails
Not Completed | 1; 7 Fingernails | 1; 2 Fingernails
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Units Other Than Participants: Fingernails
Groups:
- Platelet-rich Plasma: The proximal nail fold is cleansed with alcohol and plasma obtained from the patient is injected using a 1ml syringe and 30g needle, 0.1-0.2 ml of platelet-rich plasma is injected into the proximal nail folds.
  Blood will be drawn from a vein in the patient's arm into an 11 ml Eclipse platelet-rich plasma Tube. The blood is processed using a centrifuge machine from eclipse medical. After centrifugation, the platelet-poor portion will be separated from the platelet-rich portion.
- Platelet-poor Plasma: The proximal nail fold is cleansed with alcohol and plasma obtained from the patient is injected using a 1ml syringe and 30g needle, 0.1-0.2 ml of platelet-poor plasma is injected into the proximal nail folds.
  Blood will be drawn from a vein in the patient's arm into an 11 ml Eclipse platelet-rich plasma Tube. The blood is processed using a centrifuge machine from eclipse medical. After centrifugation, the platelet-poor portion will be separated from the platelet-rich portion
- Total: Total of all reporting groups
Arm/Group | Platelet-rich Plasma | Platelet-poor Plasma | Total
Number analyzed (Participants) | 11 | 11 | 11
Number analyzed (Fingernails) | 80 | 22 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (6) | 67.8 (6) | 67.8 (6)
Sex/Gender, Customized [Number; unit: participants]
  Female | 10 | 10 | 10
  Male | 1 | 1 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 10 | 10
  More than one race | 0 | 0 | 0
  Unknown Race or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 2 | 2 | 2
  Not Hispanic or Latino | 9 | 9 | 9
  Unknown Ethnicity or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 11
Physician Global Assessment (PGA) [Mean (Full Range); unit: score on a scale] — The Physician Global Assessment evaluates the presence and severity of five features that may occur in patients with brittle nail syndrome. Each component is scored from 0 to 3, with 3 indicating the most severe features. This results in a final score per fingernail ranging from 0 to 15. The obtained score correlates proportionally with the severity level of brittle nail syndrome.
  score on a scale | 3.16 [0 to 12] | 2.7 [0 to 10] | 3.06 [0 to 12]
Nail Superficial Abnormality Index (NSAI) [Mean (Full Range); unit: score on a scale] — The Nail Surface Abnormality Index (NSAI) assesses four parameters-pitting, discoloration, longitudinal ridging, and horizontal ridging-across four quadrants of the nail plate. Each parameter is assigned a score of 1 for presence or 0 for absence. Consequently, the highest achievable score for a nail ranges from 0 to 16, indicating the most severe abnormality.
  score on a scale | 3.5 [0 to 8] | 3.4 [0 to 8] | 3.5 [0 to 8]
Modified Nail Psoriasis Quality of Life Scale (NPQ10) [Mean (Full Range); unit: Percentage] — The modified NPQ10 comprises 10 questions gauging the impact of brittle nail syndrome on daily activities. Each response is scored from 0 to 2, resulting in a total score between 0 and 20, where higher values indicate a more significant impact. The final scores are converted to percentages, ranging from 0% to 100%, with higher percentages indicating higher functional difficulty experienced. The value reported is the average score for all study participants.
  Percentage | 16.5 [0 to 75] | 16.5 [0 to 75] | 16.5 [0 to 75]

OUTCOME MEASURES:

1. Primary Outcome: Physician Global Improvement Assessment (PGIA)
Description: The PGIA will be based on a comparison of photographs taken at baseline to the nails at week 16 of follow-up. The Physician Global Improvement Score (PGIA) evaluates the improvement of lamellar splitting, transverse splitting, ridges, longitudinal grooves, longitudinal splitting, and nail thickness in target fingernails. Change is classified as excellent, good, or fair, or categorized as no improvement or worsening.
Time Frame: At 16 weeks
Population: Per protocol population, defined as participants completing 16-week follow-up visit
Measure: Count of Units; unit: Fingernails
Units Other Than Participants: Fingernails
Arm/Group | Platelet-rich Plasma | Platelet-poor Plasma
Number analyzed (Participants) | 10 | 10
Number analyzed (Fingernails) | 73 | 20
Fingernails
  Excellent improvement | 5 | 2
  Good improvement | 7 | 1
  Fair improvement | 9 | 2
  No improvement | 42 | 13
  Worse | 10 | 2

2. Secondary Outcome: Change From Baseline in Qualify of Life, as Measured by the Modified Nail Psoriasis Quality of Life Scale (NPQ10) Between Baseline and Week 16
Description: The modified NPQ10 comprises 10 questions gauging the impact of brittle nail syndrome on daily activities. Each response is scored from 0 to 2, resulting in a total score between 0 and 20, where higher values indicate a more significant impact. The final scores are converted to percentages, ranging from 0% to 100%, with higher percentages indicating higher functional difficulty experienced. The absolute change in NPQ10 percentage score from baseline to week 16 is reported here.
Time Frame: Subjective assessments of quality of life impact due to nail health will be collected at baseline and week 16
Population: Per protocol population, defined as participants completing the 16-week follow-up visit.
Measure: Mean (Full Range); unit: percentage
Groups:
- All Groups: The proximal nail fold is cleansed with alcohol and platelet-rich plasma obtained from the patient is injected using a 1ml syringe and 30g needle, 0.1-0.2 ml of platelet-rich plasma or platelet-poor plasma is injected into the proximal nail folds.
  Blood will be drawn from a vein in the patient's arm into an 11 ml Eclipse platelet-rich plasma Tube. The blood is processed using a centrifuge machine from eclipse medical. After centrifugation, the platelet-poor portion will be separated from the platelet-rich portion.
Arm/Group | All Groups
Number analyzed (Participants) | 10
percentage | 10 [0 to 60]

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: Adverse events are reported using fingernails as unit. Adverse events were recorded for 10 subjects because one participant was lost to follow-up.
Arm/Group | Platelet-rich Plasma | Platelet-poor Plasma
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 4/10 | 4/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Platelet-rich Plasma (N=10) | Platelet-poor Plasma (N=10)
Subungual hematoma (Skin and subcutaneous tissue disorders) | 3 | 2 — Units (fingernails) affected/at risk: 3/73 in the platelet-rich plasma group 1/20 in the platelet-poor plasma group
Onychomadesis (Skin and subcutaneous tissue disorders) | 2 | 2 — Units (fingernails) affected/at risk: 4/73 in the platelet-rich plasma group 2/20 in the platelet-poor plasma group
Leukonychia (Skin and subcutaneous tissue disorders) | 1 | 0 — Units (fingernails) affected/at risk: 1/73 in the platelet-rich plasma group 0/20 in the platelet-poor plasma group
Beau's line(s) (Skin and subcutaneous tissue disorders) | 1 | 0 — Units (fingernails) affected/at risk: 1/73 in the platelet-rich plasma group 0/20 in the platelet-poor plasma group

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-14): https://cdn.clinicaltrials.gov/large-docs/07/NCT04941807/Prot_SAP_000.pdf